CLINICAL TRIAL: NCT04298697
Title: Biomarkers for Event-driven PrEP Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen Kelley, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00116781; CDC-IRB00116781 (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: Pre-exposure prophylaxis (PrEP); Post-exposure prophylaxis (PEP)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TDF/FTC for 1 week (Experimental): The first 10 participants (Arm A) will take TDF/FTC for three consecutive days of one week, taking 2 pills on the first day and one pill on the second and third day, for a total of 4 doses.
  Interventions: Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF/FTC)
- TDF/FTC for 13 weeks (Experimental): The second 10 participants (Arm B) will take TDF/FTC for three consecutive days for thirteen weeks, taking 2 pills on the first day and one pill on the second and third day of each week, for a total of 52 doses.
  Interventions: Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF/FTC)
- TDF/FTC for 13 weeks with weekly alternating schedule (Experimental): The third 10 participants (Arm C) will take TDF/FTC for three consecutive days, alternating weeks over a 13-week period, taking 2 pills on the first day and one pill on the second and third day of each dosing week, for a total of 28 doses.
  Interventions: Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF/FTC)
- TDF/FTC for 13 weeks with weekly alternating schedule every two weeks (Experimental): The fourth 10 participants (Arm D) will take TDF/FTC for three consecutive days over a 13-week period, alternating two weeks of study medication followed by two weeks with no medication, taking 2 pills on the first day and one pill on the second and third day of dosing each week, for a total of 28 doses.
  Interventions: Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF/FTC)

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) — TDF/FTC is a combination anti-HIV medication that contains the drugs tenofovir disoproxil fumarate (300 mg) and emtricitabine (200 mg). Participants will take 2 pills on the first day of the week and one pill per day on the second and third days of the week, according to the dosing schedule of the study arm they are in. Participants will have biologic specimens collected at specific time points until 28 days after the last dose.
  Other Names: Truvada

SUMMARY:
This study aims to recruit 40 participants who will take the combination anti-HIV drug tenofovir+emtricitabine (TDF/FTC) at specified times. Participants will then provide biologic samples for the measurement of anti-retroviral drug concentrations in various body compartment sites. Participants will be involved in the study for up to 24 weeks.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) continue to be disproportionately affected by HIV. In 2014, MSM made up approximately 2% of the U.S. population but accounted for 70% of the new HIV infections. The majority of MSM acquire HIV after exposure to the rectal mucosa through receptive anal intercourse without condoms. Pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP) are recommended for MSM who may be exposed to HIV to prevent infection. Current recommendations for PrEP are to take the combination anti-HIV drug, tenofovir+emtricitabine (TDF/FTC), on a daily basis for the duration of someone's HIV risk exposure period, which could be months or years. For PEP, a three-drug anti-HIV medication is recommended within 72 hours of a possible exposure for a 28-day course. While PrEP and PEP are effective, some people find it difficult to follow the recommended regimen. Therefore, additional short-course dosing regimens for PrEP and PEP are being implemented, such as on-demand or event-driven PrEP (ED-PrEP). This dosing regimen has patients take two doses of PrEP 2 to 24 hours before sex, one dose 24 hours after sex, and another dose 48 hours after sex. This study seeks to evaluate the usefulness of biomarkers to confirm self-reported adherence to ED-PrEP in MSM. The study drug provided in this study will not protect participants from HIV or treat any active infection.

This study will recruit 40 HIV-negative MSM aged 18-59 in good general health. Participants will be sequentially assigned to one of four study arms which will determine when they will take doses of the study drug and give specimen samples. All participants will provide written informed consent at the first study visit and undergo a screening medical history, physical exam, and safety laboratory tests. All participants will take at least 4 doses (pills) of the study drug. At study visits, participants will return to donate blood, hair, and urine samples, and a finger stick. All biologic specimens collected will be transferred to the Centers for Disease Control and Prevention (CDC) on the day of collection for measurement of drug levels.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative person, who was assigned male at birth, who reports sex with another man in the last year, and is in good general health.
* Not currently taking PrEP and no plans to initiate during study
* Not currently taking PEP
* Consistent condom use and willing to use condoms for the duration of the study
* Able to provide informed consent in English
* No plans for relocation in the next 4 months
* Willing to undergo peripheral blood, urine, hair, finger stick, and optional hair sampling
* Willing to use study products as directed
* Hepatitis B surface antigen (HBsAg) must be negative (screening lab test)
* Creatinine clearance (CrCl) >60 ml/min

Exclusion Criteria:

* Currently infected with hepatitis virus and/ or has liver disease
* Current or chronic history of kidney disease or CrCl<60 ml/min
* Continued need for, or use during the 90 days prior to enrollment, of the following medications:

  * Systemic immunomodulatory agents
  * Supraphysiologic doses of steroids (short course steroids less than 7 days duration, allowable at the discretion of the investigators)
  * Chemotherapy or radiation for treatment of malignancy
  * Experimental medications, vaccines, or biologicals
* Intent to use HIV antiretroviral pre/post-exposure prophylaxis (PrEP or PEP) during the study, outside of the study procedures
* Current use of hormonal therapy
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Hope Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (e.g., text, tables, figures, and appendices), will be made available for sharing.
Supporting Information: Study Protocol
Time Frame: Data will become available to researchers who provide a methodologically sound proposal, beginning 9 months and ending at 36 months following publication.
Access Criteria: Proposals should be directed to colleen.kelley@emory.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Hope Clinic in Atlanta, Georgia, USA. Participant enrollment began February 28, 2020 and all follow-up assessments were completed by August 9, 2022.
Groups:
- Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC) for 1 Week: The first 10 participants (Arm A) were assigned to take TDF/FTC for three consecutive days of one week, taking 2 pills on the first day and one pill on the second and third day, for a total of 4 doses.
  TDF/FTC is a combination anti-HIV medication that contains the drugs tenofovir disoproxil fumarate (300 mg) and emtricitabine (200 mg). Participants took 2 pills on the first day of the week and one pill per day on the second and third days of the week, according to the dosing schedule of the study arm they were in. Participants had biologic specimens collected at specific time points until 28 days after the last dose.
- TDF/FTC for 13 Weeks: The second 10 participants (Arm B) were assigned to take TDF/FTC for three consecutive days for thirteen weeks, taking 2 pills on the first day and one pill on the second and third day of each week, for a total of 52 doses.
  TDF/FTC is a combination anti-HIV medication that contains the drugs tenofovir disoproxil fumarate (300 mg) and emtricitabine (200 mg). Participants took 2 pills on the first day of the week and one pill per day on the second and third days of the week, according to the dosing schedule of the study arm they were in. Participants had biologic specimens collected at specific time points until 28 days after the last dose.
- TDF/FTC for 13 Weeks With Weekly Alternating Schedule: The third 10 participants (Arm C) were assigned to take TDF/FTC for three consecutive days, alternating weeks over a 13-week period, taking 2 pills on the first day and one pill on the second and third day of each dosing week, for a total of 28 doses.
  TDF/FTC is a combination anti-HIV medication that contains the drugs tenofovir disoproxil fumarate (300 mg) and emtricitabine (200 mg). Participants took 2 pills on the first day of the week and one pill per day on the second and third days of the week, according to the dosing schedule of the study arm they were in. Participants had biologic specimens collected at specific time points until 28 days after the last dose.
- TDF/FTC for 13 Weeks With Weekly Alternating Schedule Every Two Weeks: The fourth 10 participants (Arm D) were assigned to take TDF/FTC for three consecutive days over a 13-week period, alternating two weeks of study medication followed by two weeks with no medication, taking 2 pills on the first day and one pill on the second and third day of dosing each week, for a total of 28 doses.
  TDF/FTC is a combination anti-HIV medication that contains the drugs tenofovir disoproxil fumarate (300 mg) and emtricitabine (200 mg). Participants took 2 pills on the first day of the week and one pill per day on the second and third days of the week, according to the dosing schedule of the study arm they were in. Participants had biologic specimens collected at specific time points until 28 days after the last dose.
Period: Overall Study
Arm/Group | Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC) for 1 Week | TDF/FTC for 13 Weeks | TDF/FTC for 13 Weeks With Weekly Alternating Schedule | TDF/FTC for 13 Weeks With Weekly Alternating Schedule Every Two Weeks
Started | 15 | 17 | 6 | 5
Completed (Attended the study visit occurring 24 hours post-final dose of study medication.) | 10 | 9 | 3 | 2
Not Completed | 5 | 8 | 3 | 3
Not completed — Lost to Follow-up | 5 | 5 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- TDF/FTC for 1 Week: The first 10 participants (Arm A) were assigned to take TDF/FTC for three consecutive days of one week, taking 2 pills on the first day and one pill on the second and third day, for a total of 4 doses.
- TDF/FTC for 13 Weeks: The second 10 participants (Arm B) were assigned to take TDF/FTC for three consecutive days for thirteen weeks, taking 2 pills on the first day and one pill on the second and third day of each week, for a total of 52 doses.
- TDF/FTC for 13 Weeks With Weekly Alternating Schedule: The third 10 participants (Arm C) were assigned to take TDF/FTC for three consecutive days, alternating weeks over a 13-week period, taking 2 pills on the first day and one pill on the second and third day of each dosing week, for a total of 28 doses.
- TDF/FTC for 13 Weeks With Weekly Alternating Schedule Every Two Weeks: The fourth 10 participants (Arm D) were assigned to take TDF/FTC for three consecutive days over a 13-week period, alternating two weeks of study medication followed by two weeks with no medication, taking 2 pills on the first day and one pill on the second and third day of dosing each week, for a total of 28 doses.
- Total: Total of all reporting groups
Arm/Group | TDF/FTC for 1 Week | TDF/FTC for 13 Weeks | TDF/FTC for 13 Weeks With Weekly Alternating Schedule | TDF/FTC for 13 Weeks With Weekly Alternating Schedule Every Two Weeks | Total
Number analyzed (Participants) | 15 | 17 | 6 | 5 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 6 | 5 | 43
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (7.3) | 34.6 (9.3) | 33.2 (11.8) | 29.0 (14.2) | 32.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 15 | 17 | 6 | 5 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 0 | 1 | 7
  Not Hispanic or Latino | 12 | 14 | 6 | 4 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 2 | 2 | 17
  White | 7 | 9 | 3 | 3 | 22
  More than one race | 1 | 2 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 17 | 6 | 5 | 43

OUTCOME MEASURES:

1. Primary Outcome: Tenofovir-diphosphate (TFV-DP) Concentration
Description: Concentration of TFV-DP was measured 24 hours after the last dose to compare accumulation of drug following weekly event-driven PrEP (ED-PrEP) dosing. Dried blood spot samples were collected from participants using a 6 millimeter (mm) dried blood spot card punch system.
Time Frame: 24 Hours After Last Dose (Week 1 for Arm A, Week 13 for Arms B, C, and D)
Population: This analysis includes participants who attended the study visit that occurred 24 hours after the last dose of study medication and consistently took the study medication. Three participants in Arm B, assigned to take TDF/FTC for 13 weeks, stopped dosing early or had missed doses and were not included in this analysis since they may not have achieved steady-state drug levels as intended.
Measure: Median (Inter-Quartile Range); unit: femtomoles
Arm/Group | TDF/FTC for 1 Week | TDF/FTC for 13 Weeks | TDF/FTC for 13 Weeks With Weekly Alternating Schedule | TDF/FTC for 13 Weeks With Weekly Alternating Schedule Every Two Weeks
Number analyzed (Participants) | 10 | 6 | 3 | 2
femtomoles | 217 [154 to 267] | 1041 [540 to 1241] | 578 [450 to 1240] | 789 [261 to 1317]

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning when individuals gave consent to participate in the study and continued through the final assessment, for up to a total of 24 weeks.
Arm/Group | TDF/FTC for 1 Week | TDF/FTC for 13 Weeks | TDF/FTC for 13 Weeks With Weekly Alternating Schedule | TDF/FTC for 13 Weeks With Weekly Alternating Schedule Every Two Weeks
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT04298697/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT04298697/ICF_001.pdf